CLINICAL TRIAL: NCT00537264
Title: A Randomized Controlled Trial Comparing Computer- Versus Interviewer-administered Approach for Assessing Health-related Quality of Life in Multi-Ethnic Singapore
Brief Title: A Comparison of Computerised Versus Interviewer-administered Approach for Assessing Health-related Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 03/1/27/18/226
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Diabetes; Heart Disease; Hypertension; Stroke
Keywords: health-related quality of life; primary care; computer-assisted instruction
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Hypertension; Stroke | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer (Experimental): Health-related quality of life questionnaires will be administered using a computerised multimedia touchscreen system.
  Interventions: Other: Health-related quality of life assessment
- Interviewer (Experimental): Health-related quality of life questionnaire will be administered via face-to-face interviews.
  Interventions: Other: Health-related quality of life assessment

INTERVENTIONS:
Other: Health-related quality of life assessment — Study participants will be asked to complete the following health-related quality of life questionnaires: EQ-5D, Health Utilities Index 3, SF-8 and SF-6D. The Singapore (Chinese) versions of these questionnaires have been previously tested and validated in a pilot cohort of the same study population.
  Other Names: Patient-reported outcomes
  Arms: Computer
Other: Health-related quality of life assessment — Study participants will be asked to complete the following health-related quality of life questionnaires: EQ-5D, Health Utilities Index 3, SF-8 and SF-6D. The Singapore (Chinese) versions of these questionnaires have been previously tested and validated in a pilot cohort of the same study population.
  Other Names: Patient-reported outcomes
  Arms: Interviewer

SUMMARY:
The aim of this study is to compare a multimedia, computerised approach vs. interviewer administration of health-related quality of life (HRQoL) instruments.

DETAILED DESCRIPTION:
There are no drug treatments involved in this study. The administration of health-related quality of life questionnaires is the intervention being studied. Health-related quality of life questionnaires measure the physical, mental and social well-being of an individual, are recognised as important patient-reported outcomes and are increasingly being used in clinical trials and routine clinical practice. By asking study participants to complete a questionnaire assessing their physical, mental and social well-being, we are increasing their awareness of these aspects of their health and may directly or indirectly prompt them to take actions and/ or have thoughts that may improve or worsen their health status. Hence, we have considered this an interventional study. This survey will be conducted in Chinese.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 and above
* Singaporean citizens or permanent residents
* Speaks Mandarin

Exclusion Criteria:

* Patients who are mentally incapable of completing a questionnaire

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life outcomes | Past 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julian Thumboo, FRCP (Edin), Principal Investigator — Singapore General Hospital
Locations (1):
- Geylang Polyclinic, 21 Geylang East Central, Singapore, Singapore

REFERENCES:
- [Background] Thumboo J, Wee HL, Cheung YB, Machin D, Luo N, Fong KY. Development of a Smiling Touchscreen multimedia program for HRQoL assessment in subjects with varying levels of literacy. Value Health. 2006 Sep-Oct;9(5):312-9. doi: 10.1111/j.1524-4733.2006.00120.x. PMID 16961549